CLINICAL TRIAL: NCT02300922
Title: Pretargeted Radioimmunotherapy in Metastatic Colorectal Cancer : A Multicentric Phase I/II Study of Fractionated TF2 Plus 90Y-IMP288 (RITCOLON)
Brief Title: Pretargeted Radioimmunotherapy in Metastatic Colorectal Cancer
Acronym: RITCOLON
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Premature termination of recruitment due to the discontinuation of product supply by the project's industrial partner.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC14_0003
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- several cohorts (Experimental): All patients will receive 3 injections of TF2 (the first: 14 mg/m², the second and the third:75 mg/m²). One day after each injection of TF2, the patient will receive a radiolabelled peptide (IMP-288) with Yttrium for therapeutic injectionThe First cohort will receive 555 MBq/m2 X 2 of 90-Y-IMP-288.:
  All patient will receive 180 MBq of 111-In-IMP-288 for dosimetry analysis
  Interventions: Drug: Antibody TF2; Drug: 90-Y-IMP-288; Drug: 111-In-IMP-288

INTERVENTIONS:
Drug: Antibody TF2 — injection of a recombinant antibody CEA specific. Three injections. Each injection are separate by one week
Drug: 90-Y-IMP-288 — Injection of the peptide 90-Y-IMP-288, 24 Hours after injection of TF2. 2 injections by patients separated by one week (week 2 and week 3)
Drug: 111-In-IMP-288 — Injection of the peptide 111-In-IMP-288, 24 Hours after the first injection of TF2 (week 1)

SUMMARY:
Phase I/II, Open-labeled, Prospective, Multi-center study of a Pretargeted Radioimmunotherapy in metastatic colorectal cancer with ractionated injections of TF2 plus 90Y-IMP288 (RITCOLON).

DETAILED DESCRIPTION:
This study investigates a pretargeted radioimmunotherapy (pRAIT) with the anti-carcinoembryonic antigen (CEA) TF2 bispecific monoclonal antibody (BsMAb) and the 90Y-IMP288 radio-labeled peptide.

TF2 will be given once a week for 3 successive weeks at 75 mg/m2 per dose. IMP288 will be given 3 times, 1 day after each TF2 injection. IMP288 will be radio-labeled with 111In (imaging) for the first injection and then 90Y (therapy) for the 2 subsequent injections.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic colorectal cancer and failure to standard therapies (5-fluorouracil, irinotecan, oxaliplatin, anti-vascular endothelium growth factor, anti-epidermal growth factors in patients with RAS wild type tumors). A previous line with regorafenib is not required.
2. Elevated CEA serum level or proved CEA expression in tumor tissue
3. ≥ 18 years of age,
4. Given signed, written informed consent
5. Existence of at least one measurable tumor lesion by CT or MRI at the time of treatment, but no single lesion ≥ 8 cm in diameter.
6. At least 4 weeks recovery period after any major surgery, radiation, or chemotherapy, and total recovery from any acute toxicities associated with these prior treatments.
7. Life expectancy ≥ 3 months, Karnofsky performance status of ≥ 70%
8. Adequate hematology and renal function and hepatic function
9. Patients of childbearing potential must be willing to practice birth control during the study until at least 12 weeks after treatment, and women of childbearing potential must have a negative serum pregnancy test to enter the study

Exclusion Criteria :

1. Known central nervous system metastatic disease
2. > 25% bone marrow involvement
3. CEA plasma levels >2,000 ng/mL
4. Patients with successfully treated non-melanoma skin cancer or carcinoma in situ of the cervix are eligible, while patients with other prior malignancies must have had at least a 3-year disease-free interval.
5. HIV positive, hepatitis B-antigen positive, or hepatitis C positive patients
6. Known autoimmune disease,
7. Known history of unstable angina, myocardial infarction, or congestive heart failure present within 6 months or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy, no known history of clinical significant, active chronic obstructive pulmonary disease, or other moderate to severe chronic respiratory illness present within 6 months
8. Infection requiring intravenous antibiotic use within 1 week before inclusion,
9. Corticosteroids are not allowed within 2 weeks of study entry nor during the study except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis.
10. Patients who received a treatment containing a nitrosourea compound will not be enrolled for at least 6 weeks after the end of that treatment.
11. Known hypersensitivity to murine antibodies or proteins
12. Immunization against TF2 for patients who has already received injection of TF2
13. Adult patient unable to give informed consent because of intellectual impairment.
14. Adult patient protected by the French law

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose for 90Y-IMP288. | Week 6 to week 12
  toxicity analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France